CLINICAL TRIAL: NCT02470078
Title: Randomised Controlled Trial of Pharyngeal Electrical Stimulation for the Treatment of Post-extubation Dysphagia in Acute Stroke Patients
Brief Title: Pharyngeal Electrical Stimulation for the Treatment of Post-extubation Dysphagia in Acute Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014-155
Record Dates: First submitted 2015-06-03; First posted 2015-06-12 (Estimated); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Stroke; Dysphagia
Keywords: extubation
MeSH Terms: conditions — Stroke; Deglutition Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Pharyngeal electrical stimulation (Experimental): Pharyngeal electrical stimulation once daily for 10 minutes on three consecutive days.
  Interventions: Device: Phagenyx-Catheter, Phagenesis Limited, UK.
- Sham stimulation (Sham Comparator): Sham stimulation once daily for 10 minutes on three consecutive days.
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Phagenyx-Catheter, Phagenesis Limited, UK. — Pharyngeal electrical stimulation via an intraluminal catheter (Phagenesis Ltd.) once daily for 10 minutes on three consecutive days. The intensity of the electrical stimulation is determined following the calculation of suitable sensory threshold, tailored to the individual patients. After determining the optimal stimulation intensity, 10 minutes of stimulation are delivered.
  Arms: Pharyngeal electrical stimulation
Device: Sham stimulation — The intraluminal catheter (Phagenesis Ltd.) for pharyngeal electrical stimulation is placed. In the sham group the optimisation procedure was imitated as closely as possible to mitigate any bias or effect of time spent interacting with the patient during PES, but no current was applied. After this procedure 10 min of sham stimulation were delivered.
  Arms: Sham stimulation

SUMMARY:
The purpose of this study is to evaluate whether pharyngeal electrical stimulation in addition to standard care can enhance swallowing recovery in severely dysphagic stroke patients post extubation compared to sham treatment plus standard care.

ELIGIBILITY:
Inclusion Criteria:

- severe dysphagia post extubation due to acute stroke

Exclusion Criteria:

* preexisting dysphagia
* comorbidities that can possibly cause dysphagia
* psychiatric comorbidities
* pacemaker or other implanted electronic devices

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Reintubation rate | 120 hours
  Need for reintubation within 120 hours from extubation
Pneumonia rate | 120 hours
  Incidence of aspiration pneumonia within 120 hours from extubation

SECONDARY OUTCOMES:
Length of stay | Participants will be followed for the duration of stay on the intensive care unit, an expected average of 3 weeks
  Length of stay on the intensive care unit
Time until oral nutrition | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  Time span from extubation until consumption of an completely oral diet is safely possible
PEG tube placement | Participants will be followed for the duration of hospital stay, an expected average of 5 weeks.
  Number of participants needing percutaneous endogastric tube placement due to persistent severe dysphagia
Swallowing function | after 3 days of treatment
  Salient semiquantitative parameters of swallowing function (leaking, penetration, aspiration, residues, delayed triggering of swallow reflex) as assessed by a standardized fiberoptic endoscopic evaluation protocol after three days of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Dziewas, MD, Principal Investigator — University Hospital Münster
Locations (1):
- Department of Neurology, University of Muenster, Münster, Germany

REFERENCES:
- [Derived] Suntrup-Krueger S, Labeit B, Marian T, Schroder J, Claus I, Ahring S, Warnecke T, Dziewas R, Muhle P. Pharyngeal electrical stimulation for postextubation dysphagia in acute stroke: a randomized controlled pilot trial. Crit Care. 2023 Oct 3;27(1):383. doi: 10.1186/s13054-023-04665-6. No abstract available. PMID 37789340